CLINICAL TRIAL: NCT01169688
Title: Preoperative Cataract Pupillary Dilation: Inpatient vs Outpatient
Brief Title: Preoperative Cataract Pupillary Dilation: Inpatient At The Ambulatory Surgery Center vs Outpatient Dilation Prior To Arrival At The Ambulatory Surgery Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Kansas Surgery Center (Other)
Responsible Party: Ronald Holweger MD, Northwest Kansas Surgery Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NWKSC_2007_01
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2007-12

CONDITIONS: Pupil Dilation Prior to Cataract Surgery In-patient; Pupil Dilation Prior to Cataract Surgery Out-patient
Keywords: Cataract Surgery; Pupillary Dilation
MeSH Terms: conditions — Mydriasis | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pupil dilation with phenylephrine 10% vs cyclopentolate 2%

SUMMARY:
This study was done to compare efficacy, safety and efficiencies of various methods of pupil dilation prior to cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to self administer eye or have a helper for the task of administering eye drops.
* Ability to follow and eye drop administration schedule.
* No noted ocular abnormalities.
* Bilateral cataract surgery anticipated.

Exclusion Criteria:

* Inability to self administer eye drops or have assistance with eye drop administration.
* Health problems that would contraindicate self administration of dilating eye drops such as poor cardiovascular or respiratory status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)